CLINICAL TRIAL: NCT03984955
Title: A Prospective, Double Blind, Single Centre, RCT, Comparing the Effectiveness of Physiotherapy in Addition to One of 3 Types of Image Guided Injection of the Common Extensor Tendon, on Pain and Function in Patients With Tennis Elbow.
Brief Title: Comparing Injection Treatments for Tennis Elbow
Acronym: CITTE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wrightington, Wigan and Leigh NHS Foundation Trust (Other)
Collaborators: TRB Chemedica (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R&D 1026
Record Dates: First submitted 2019-02-21; First posted 2019-06-13 (Actual); Last update posted 2024-08-06 (Actual); Status verified 2024-08

CONDITIONS: Tennis Elbow; Lateral Epicondylitis; Elbows Tendonitis
MeSH Terms: conditions — Tennis Elbow

STUDY DESIGN:
Intervention Model Description: Prospective, Controlled, Randomised, Double Blind, Single Centre Trial
Who Masked: Participant, Outcomes Assessor
Masking Description: The patient will be blinded/masked to their group allocation: For Groups (B) and (C), the withdrawn blood will be discarded into a suitable clinical waste container out of sight of the participant in an adjoining room. The centrifuge, also in the adjoining room, will be set to run at 32000rpm for 15 minutes in order to aid in participant blinding.
  The class-based physiotherapy sessions will be taught be a physiotherapist who is blind to the treatment allocation of the study participants attending the class.
  The outcome assessments will be recorded by a member of the research team blind to the participant's treatment allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group A PRP injection (Active Comparator): Platelet-Rich Plasma injection Single therapeutic injection of Platelet-Rich Plasma performed under ultrasound guidance.
  This group will also undergo a class-based physiotherapy intervention. This outcomes for this group will be compared to those receiving Sodium hyaluronate with mannitol (Ostenil Tendon) and those receiving the sham injection.
  Interventions: Device: Platelet-Rich Plasma Injection
- Group B Ostenil Tendon (Active Comparator): Sodium hyaluronate with mannitol (Ostenil Tendon) Single therapeutic injection of sodium hyaluronate with mannitol (marketed under the device name Ostenil Tendon) under ultrasound guidance. This group will also undergo a class-based physiotherapy intervention.
  Interventions: Device: Sodium hyaluronate with mannitol (Ostenil Tendon)
- Group C control group (Sham Comparator): Subcutaneous sham injection. This group will also undergo a class-based physiotherapy intervention. The outcomes for this group will be compared to those receiving Sodium hyaluronate with mannitol (Ostenil Tendon) and to those receiving PRP injection.
  Interventions: Other: Subcutaneous sham injection

INTERVENTIONS:
Device: Sodium hyaluronate with mannitol (Ostenil Tendon) — 1ml isotonic solution contains 20.0mg sodium hyaluronate and sodium chloride, disodium phosphate, sodium dihydrogen phosphate, mannitol and water for injections.
  Other Names: Ostenil Tendon
  Arms: Group B Ostenil Tendon
Device: Platelet-Rich Plasma Injection — Platelet-rich plasma (PRP) describes an autologous blood plasma fraction enriched with platelets which is then injected at the site of tendon injury.
  Arms: Group A PRP injection
Other: Subcutaneous sham injection — Sham injection will penetrate the skin, but no therapeutic substance will be injected
  Arms: Group C control group

SUMMARY:
Tennis elbow is one of the most common musculoskeletal problems affecting the arm and is thought to be mainly due to overuse of the muscles that extend the wrist. The pain arises from the lateral epicondyle of the humerus, where the tendons of the wrist extensor muscles attach.

There are many treatment options available for tennis elbow including oral medication, physiotherapy and injection therapy. Surgical options are reserved for those who fail to respond to more conservative treatments. Physiotherapy is a widely used, non-invasive treatment option for the management of tennis elbow. Research has shown that in the longer term, physiotherapy is superior to corticosteroid injection in the treatment of tennis elbow and a meta-analysis of published research concluded that Platelet Rich Plasma injection and Hyaluronic Acid injection are superior to corticosteroid for long term pain relief in tennis elbow.

At present there is not enough evidence to indicate what the 'Gold Standard' treatment for tennis elbow is, and more research is therefore needed to help guide decision-making. The aim of this study is therefore to examine the effects of injection therapy in addition to physiotherapy treatment, in comparison to physiotherapy and a control injection on pain and function in patients with tennis elbow.

All participants in this study will undergo a structured, specifically designed, class-based physiotherapy intervention, in addition to being randomly allocated to receive one of the following three types of injection: (a) a control injection whereby a needle is inserted into the skin but no therapeutic substance is injection, (b) a single therapeutic injection of platelet-rich plasm or (c) a single therapeutic injection of hyaluronic acid. Baseline data will be collected at the time of recruitment and participants will be followed up at 3 months and 12 months post treatment. Outcomes will be assessed using various patient-reported outcome measures in addition to clinical examination. The primary outcome for this study is the improvement in the quick DASH score at 12 months post-treatment compared to baseline.

DETAILED DESCRIPTION:
The design of the current study is a prospective, randomised, controlled, double blinded, single centre trial.

On the day of their initial appointment in the outpatient department, patients diagnosed with tennis elbow by their consultant who meet all of the necessary inclusion and exclusion criteria will be introduced to the study by the consultant. They will also be provided with a copy of the participant information sheet.

When the potential participant then attends their pre-operative assessment appointment, they will be invited to discuss the study further with a member of the host Trust's research team. If they then wish to proceed, they will be invited to read and sign a copy of the study consent form. Consenting patients will then be asked to complete a questionnaire designed to record all relevant demographic data including: Age, gender, affected side, dominant side, weight, height (so that BMI may be calculated), duration of symptoms, current use of pain-relieving medications, occupation, leisure activities and ethnicity. They will also be asked to complete a visual analogue pain scale, and the following 4 validated patient reported outcome measures.

Following completion of the patient reported outcome questionnaires, participants will then be randomised to one of the following three treatment groups: Group(A)will receive a standardised, class-based physiotherapy program in addition to a single therapeutic injection of Platelet-Rich Plasma; Group (B) will undergo an identical physiotherapy program to group A, but with a single therapeutic injection of sodium hyaluronate with mannitol; or group (C) who will undergo an identical physiotherapy program to both groups (A) and (B), however they will receive a sham injection, which will penetrate the skin, but no therapeutic substance will be injected.

The randomisation sequence will be generated using freely available online randomisation facilities prior to the start of the study. Participants will be randomised to either Group A, Group B or Group C in a 1:1:1 ratio (see above for group descriptions). The allocation sequence will be concealed in sealed opaque envelopes which will be prepared prior to the start of the study and will be opened after informed consent has been gained and baseline data has been collected.

Consenting participants will all attend Wrightington Hospital for their allocated injection to be administered under ultrasound guidance to ensure accurate needle placement. All participants will have 30mls of whole blood drawn under aseptic conditions in order to aid blinding of participants to their treatment allocation.

For those allocated to receive a PRP injection (Group A), the whole blood will be placed in a cell separator and centrifuged at 32000 rpm for 15 minutes. Whilst the blood is being centrifuged, 2ml of 2% plain lidocaine will be injected into the subcutaneus layer at the site where the PRP is to be injected. 1ml of the PRP produced will then be drawn into a syringe which will be wrapped in silver foil so as to conceal the contents from the participants. The PRP will then be injected into the lateral epicondyle via a blue (20 gauge) hypodermic needle using a peppering technique under ultrasound control.

For Groups (B) and (C), the withdrawn blood will be discarded into a suitable clinical waste container out of sight of the participant in an adjoining room. The centrifuge, also in the adjoining room, will be set to run at 32000rpm for 15 minutes in order to aid in participant blinding. For those in group (B), whilst the centrifuge is running, 2ml of 2% plain lidocaine will be injected into the subcutaneous layer at the site of injection. A pre-prepared 'Ostenil Tendon' syringe will be wrapped in silver foil (again to help conceal the nature of the contents from the participants) and 2ml will be injected into the peri-tendinous area via a blue (20 gauge) hypodermic needle under ultrasound control.

For those in group (C) whilst the centrifuge is running, 2ml of 2% plain lidocaine will be injected into the subcutaneous layer at the site of injection. An empty syringe wrapped in silver foil with a blue (20 gauge) will then be used to perform a sham injection into the subcutaneous tissue only, by passing the needles into the tissue with no injectate.

In order to further aid blinding of participants, during the procedure they will be distracted by asking them to confirm their personal details.

In order to gain a measure of how the participant's pain changes in the days and weeks following surgery, they will be given a pain diary on the day of their treatment to complete on days 1,2,3,7,14, and at 6 and 12 weeks.

Prior to discharge from the hospital participants will be taught basic home exercises by a physiotherapist who is unaware of the participant's group allocation. they will then begin a specifically designed, formal, class-based physiotherapy program 5-15 days post-injection. Exercises taught on the day of treatment will include eccentric loading exercises of the wrist extensors and they will be asked to commence these exercises the day after the injection and to complete 3 sets of 15 repetitions 3 times per day. They will also be taught simple stretches of the wrist extensors to complete after each set of eccentric strengthening exercises.

The formal physiotherapy program will include fortnightly physiotherapy classes taught by a blinded physiotherapist. After being taught the exercises on a 1:1 basis in order to ensure correct technique, the participants will be supervised during a circuit style exercise program. The circuit will include exercises to load the common extensors, strengthening of the rotator cuff muscles, strengthening of the scapular stabilising muscles and upper limb strengthening using the full kinetic chain. Participants will also be taught a home exercise program which will reflect the content of the class circuit.

At 3 months and 12 months post-injection participants will be assessed by a clinician who again is unaware of the participant's grouping. At each follow-up, the participants will be asked to complete the patient reported outcome questionnaires. They will also be asked regarding their use of rescue medication (i.e. how much analgesic medication they require to manage their pain) and this will be recorded by the clinician.

If any participant is unable to attend the hospital for follow-up at either the 3 or 12 month time-point, they will be contacted by telephone to gather the outcome information. All participants will be discharged from the care of the treating consultant at 12 weeks unless enduring or subsequently manifesting symptoms are present and the final 12 month visit will therefore be solely for the purposes of research.

ELIGIBILITY:
Inclusion Criteria:

Invitations to participate in the study will be extended to male and female patients, 18 years and above, referred to the Orthopaedic Departments who receive a diagnosis of Lateral Epicondyle Tendinosis (with or without degenerative changes) with symptoms present for > 3 months, whose symptoms and clinical evaluation warrant the prescription of a peri-tendinous injection to relieve symptoms and who are competent to give informed consent.

Exclusion Criteria:

* Absence of tenderness at the lateral epicondyle.
* Congenital or traumatic bio-mechanical deformities of Elbow complex.
* Previous Corticosteroidal, Local Anaesthetic, PRP or Hyaluronic Acid injections to target elbow within the last three months.
* Known hypersensitivity to PRP, Hyaluronic acid or any excipients associated with any of the prescribed injections.
* Known contraindication to any treatments constituting normal/appropriate therapy in the view of the Consulting clinician including local infection
* Ipsilateral arm pathology severe enough to cause confusion of localised pain perception.
* Pregnant or lactating women
* Pain score less than 4/10
* Patients commenced on medication for the treatment of anxiety or depression within the last 6 weeks
* Previous involved in research in last 12 months
* Any progressive, degenerative neuromuscular disorder

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 123 (Estimated)
Dates: Start 2018-04-18 (Actual); Primary Completion 2026-02-06 (Estimated); Study Completion 2026-02-06 (Estimated)

PRIMARY OUTCOMES:
The change in Objective functional assessment as evidenced by the change in Quick Disabilities of the Arm, Shoulder and Hand (DASH) scores from pre-treatment to 12 months post treatment. | The QuickDASH scores will be recorded at baseline, and will be repeated at 3 months and 12 months post-injection.
  The QuickDASH consists of 11 items which were extracted from the original 30-item DASH scale. To calculate a QuickDASH score, at least 10 of the 11 items must be completed. Similar to the original DASH, each item has 5 response options and, from the item scores, scale scores are calculated, ranging from 0 (no disability) to 100 (most severe disability).

SECONDARY OUTCOMES:
The change from baseline in objective pain scores as evidenced by the Visual Analogue Pain Scale (VAS) at 12 months post-treatment. | The VAS will be recorded at baseline, and will be repeated at 3 months and 12 months post-injection.
  The Visual Analogue Pain scale is a horizontal line, 100 mm in length, anchored by descriptors at each end, namely 'No pain at all' on the left side and 'Worst imaginable pain' on the right side. The patient marks on the line the point that they feel represents their perception of their current pain. The VAS score is determined by measuring in millimetres from the left hand end of the line to the point that the patient marks.
The change in objective functional assessment as evidenced by the Oxford Elbow Score (OES) | The OES will be recorded at baseline, and will be repeated at 3 months and 12 months post-injection.
  The Oxford Elbow Score (OES) is a short 12-item patient-reported outcome measure originally designed and developed for assessing outcomes of elbow surgery.The OES has 12 items (questions) with 5 response options each. Each item response is scored as 0 to 4, with 0 representing greater severity. Underlying the 12 items are 3 domains (subscales): elbow pain, elbow function and social-psychological effects. Scores for each domain are calculated as the sum of each individual item score within that domain. This gives a score range of 0-16 for each domain and 0-48 overall, with 0 indicating the worst elbow score and 48 as a 'normal' elbow score.
Change in general health-related quality of life as evidenced by change in the EQ-5D general health questionnaire. | The EQ-5D will be recorded at baseline, and will be repeated at 3 months and 12 months post-injection.
  The EQ-5D is a standardised instrument for use as a measure of health outcome. Applicable to a wide range of health conditions and treatments, it provides a simple descriptive profile and a single index value for health status. The EQ-5D descriptive system comprises the following 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 3 levels: no problems, some problems, extreme problems. The respondent is asked to indicate his/her health state by marking the box against the most appropriate statement in each of the 5 dimensions.The EQ VAS then records the respondent's self-rated health on a vertical, visual analogue scale where the endpoints are labelled 'Best imaginable health state' and 'Worst imaginable health state'. This information can be used as a quantitative measure of health outcome as judged by the individual respondents.
Relationship of pre-injection Hospital Anxiety and Depression Scale (HADS) score to the outcome | The HAD score will be recorded at baseline, and will be repeated at 3 months and 12 months post-injection.
  The Hospital Anxiety and Depression Scale (HADS) is a valid and reliable self-rating scale that measures anxiety and depression in both hospital and community settings. The HADS comprises 14 questions, seven relating to anxiety and seven relating to depression. Each item is scored from 0-3, with higher scores indicating higher symptoms frequencies. Scores for each subscale (anxiety and depression) range from 0 to 21 with scores categorized as follows: normal 0-7, mild 8-10, moderate 11-14, and severe 15-21. Scores for the entire scale (emotional distress) range from 0 to 42, with higher scores indicating more distress. Prior to completing the scale patients are asked to ensure the answers they given reflect how they have been feeling during the past week.
Change in HADS score at 12 months compared to baseline | The HAD score will be recorded at baseline, and will be repeated at 3 months and 12 months post-injection.
  See above

CONTACTS AND LOCATIONS:
Overall Officials: Adam Watts, Principal Investigator — Wrightington, Wigan and Leigh NHS Foundation Trust
Locations (1):
- Wrightington Wigan and Leigh NHS Foundation Trust, Wigan, Lancashire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gliedt JA, Daniels CJ. Chiropractic treatment of lateral epicondylitis: a case report utilizing active release techniques. J Chiropr Med. 2014 Jun;13(2):104-9. doi: 10.1016/j.jcm.2014.06.009. PMID 25685118
- [Background] Smidt N, van der Windt DA, Assendelft WJ, Deville WL, Korthals-de Bos IB, Bouter LM. Corticosteroid injections, physiotherapy, or a wait-and-see policy for lateral epicondylitis: a randomised controlled trial. Lancet. 2002 Feb 23;359(9307):657-62. doi: 10.1016/S0140-6736(02)07811-X. PMID 11879861
- [Background] Lo MY, Safran MR. Surgical treatment of lateral epicondylitis: a systematic review. Clin Orthop Relat Res. 2007 Oct;463:98-106. doi: 10.1097/BLO.0b013e3181483dc4. PMID 17632419
- [Background] Johnson GW, Cadwallader K, Scheffel SB, Epperly TD. Treatment of lateral epicondylitis. Am Fam Physician. 2007 Sep 15;76(6):843-8. PMID 17910298
- [Background] Green S, Buchbinder R, Barnsley L, Hall S, White M, Smidt N, Assendelft W. Non-steroidal anti-inflammatory drugs (NSAIDs) for treating lateral elbow pain in adults. Cochrane Database Syst Rev. 2002;(2):CD003686. doi: 10.1002/14651858.CD003686. PMID 12076503
- [Background] Beard JM, Safranek SM, Spogen D. Clinical inquiries. What treatment works best for tennis elbow? J Fam Pract. 2009 Mar;58(3):159-61. No abstract available. PMID 19284945
- [Background] Assendelft W, Green S, Buchbinder R, Struijs P, Smidt N. Tennis elbow. BMJ. 2003 Aug 9;327(7410):329. doi: 10.1136/bmj.327.7410.329. No abstract available. PMID 12907489
- [Background] Saito S, Furuya T, Kotake S. Therapeutic effects of hyaluronate injections in patients with chronic painful shoulder: a meta-analysis of randomized controlled trials. Arthritis Care Res (Hoboken). 2010 Jul;62(7):1009-18. doi: 10.1002/acr.20174. PMID 20235211
- [Background] Funk L. (2005) Hyaluronan vs Corticosteroids for Subacromial Impingement of the Shoulder. Osteoarthritis & Cartilage. 13(Suppl A)
- [Background] Petrella RJ, Cogliano A, Decaria J, Mohamed N, Lee R. Management of Tennis Elbow with sodium hyaluronate periarticular injections. Sports Med Arthrosc Rehabil Ther Technol. 2010 Feb 2;2:4. doi: 10.1186/1758-2555-2-4. PMID 20205851
- [Background] Mishra A, Pavelko T. Treatment of chronic elbow tendinosis with buffered platelet-rich plasma. Am J Sports Med. 2006 Nov;34(11):1774-8. doi: 10.1177/0363546506288850. Epub 2006 May 30. PMID 16735582
- [Derived] Karjalainen TV, Silagy M, O'Bryan E, Johnston RV, Cyril S, Buchbinder R. Autologous blood and platelet-rich plasma injection therapy for lateral elbow pain. Cochrane Database Syst Rev. 2021 Sep 30;9(9):CD010951. doi: 10.1002/14651858.CD010951.pub2. PMID 34590307

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-23): https://cdn.clinicaltrials.gov/large-docs/55/NCT03984955/Prot_SAP_000.pdf